CLINICAL TRIAL: NCT04491565
Title: An Interactive Video Educational Tool Improves the Quality of Bowel Preparation for Colonoscopy: A Randomized Controlled Trial
Brief Title: An Interactive Video Educational Tool Improves the Quality of Bowel Preparation for Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Dayna Early, Principle Investigator, Professor of Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 201909053
Record Dates: First submitted 2020-07-24; First posted 2020-07-29 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Colon Cancer Screening
Keywords: colonoscopy

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard education (No Intervention)
- educational video (Active Comparator)
  Interventions: Other: educational video

INTERVENTIONS:
Other: educational video — an interactive educational video was viewed by participants in the intervention arm.
  Arms: educational video

SUMMARY:
The investigators aimed to determine whether an interactive, online educational platform could improve procedure show rates and bowel preparation scores in an outpatient population presenting for routine colonoscopy.

DETAILED DESCRIPTION:
The investigators performed a prospective, endoscopist-blinded, randomized controlled trial at a hospital-based outpatient endoscopy center. Eligible patients were randomized to two groups. Both groups received verbal and written instructions per standard care, while the intervention group received access to an interactive, on-line video. Primary outcomes were bowel preparation scores graded using the Boston Bowel Prep Score (BBPS), procedure show rates, patient satisfaction, and pre-procedure anxiety. Secondary outcomes included adenoma detection rate, mean bowel prep score per colonic segment, total number of polyps detected, and complication rates.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Access to text messaging and the internet (mobile phone access alone was considered sufficient)
* Prescribed standard split-dose bowel preparation
* Able to provide informed consent via telephone.

Exclusion Criteria:

* Pregnant
* Mentally impaired
* Undergoing screening or surveillance for inflammatory bowel disease .

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Adequacy of bowel prep | intra procedure
  adequacy of colonoscopy bowel prep was scored from 0 (worst) to 9 (best).

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States